CLINICAL TRIAL: NCT03183193
Title: Non-alcoholic Fatty Liver Disease (NAFLD) in Overweight and Obese People Under Nutritional and Lifestyle Follow-up: a Randomized Controlled Trial
Brief Title: Fatty Liver in Obesity: Long-lifestyle Follow-up (FLiO)
Acronym: FLiO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Collaborators: Complejo Hospitalario de Navarra (Other)
Responsible Party: Principal Investigator, Marian Zulet, Principal Investigator, University of Navarra
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FLiO
Record Dates: First submitted 2017-03-31; First posted 2017-06-12 (Actual); Last update posted 2017-06-12 (Actual); Status verified 2017-06

CONDITIONS: Non-Alcoholic Fatty Liver Disease; Obese; Overweight
Keywords: NAFLD; NASH; Obesity; AASLD; AHA; Energy-restricted diet; Lifestyle intervention; Mediterranean diet; Weight loss; Liver damage; Inflammation; Oxidative stress; Microbiota composition; Eating behaviour; Satiety; Physical activity; Sedentary behaviours; Sleep quality; Sleep duration; Psychological factors; Nutrigenomics; Nutrigenetics; Transcriptomics; Epigenetics; Metabolomics; miRNAs; Lipidomics
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Obesity; Overweight; Weight Loss; Inflammation; Feeding Behavior; Motor Activity; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: The participants are randomly assigned to Control or FLiO strategy.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control diet (Placebo Comparator): A conventional and balanced diet based on American Heart Association (AHA) guidelines and lifestyle advice to achieve the objective of American Association for the Study of Liver Diseases (AASLD): loss of at least 3-5% of the initial body weight and up to 10% needed to improve necroinflammation.
  Interventions: Other: Control diet
- FLiO diet (Experimental): A mediterranean dietary strategy based on macronutrient distribution (quantity and quality), antioxidant capacity, meal frequency, dietary behaviour and lifestyle advice to achieve the objective of AASLD: loss of at least 3-5% of the initial body weight and up to 10% needed to improve necroinflammation.
  Interventions: Other: FLiO diet

INTERVENTIONS:
Other: Control diet — The participants follow a conventional and balanced distribution of macronutrients (30% fat, 15% protein, 55% carbohydrates), adequate fiber (25-30 g/day) and dietary cholesterol (<250 mg/day) intake according to AHA guidelines. This strategy was included within a personalized energy-restricted diet (-30% individual needs) under healthy lifestyle advice in order to achieve the objectives of AASLD (loss of at least 3-5% of the initial body weight and up to 10% needed to improve necroinflammation).
  Other Names: American Heart Association diet
  Arms: Control diet
Other: FLiO diet — The participants follow a strategy based on a distribution of macronutrients 30-35% lipid (extra virgin olive oil and fatty acids Ω3 in detriment of saturated, trans and cholesterol)/ protein 25% (vegetable against animal)/carbohydrates 40-45% (low glycaemic index, fiber 30-35 g/day); high adherence to the Mediterranean diet and natural antioxidants; meal frequency of 7 meals/day; size/composition of the ration suitable for each moment; including traditional foods with no additional economic cost that will allow diet adherence without abandonment; avoid inappropriate mealtimes and the eating manners as the eating rate. The participants are instructed to follow this strategy within a personalized energy-restricted diet (-30%) and under healthy lifestyle advice to achieve AASLD objectives.
  Other Names: Fatty Liver in Obesity diet
  Arms: FLiO diet

SUMMARY:
Non-alcoholic fatty liver disease (NAFLD) is a condition of excessive hepatic lipid accumulation in subjects that consume less than 20g ethanol per day, without other known causes as drugs consumption or toxins exposure. In Western countries, the rate of this disease lies about 30% in the general adult population. The process of developing NAFLD can start from simple steatosis to non-alcoholic steatohepatitis (NASH), which eventually can lead to cirrhosis and hepatocellular carcinoma in the absence of alcohol abuse. Liver biopsy is considered the "gold standard" of steatosis, fibrosis and cirrhosis. However, it is rarely performed because it is an invasive procedure and investigators are focusing in the application of non-invasive liver damage scores for diagnosis.

The pathogenesis of NAFLD is multifactorial and triggered by environmental factors such as unbalanced diets and overnutrition as well as by lack of physical activity in the context of a genetic predisposition. Nowadays, the treatment of NAFLD is based on diet and lifestyle modifications. Weight loss, exercise and healthy eating habits are the main tools to fight NAFLD. Nevertheless, there is no a well characterized dietary pattern and further studies are necessary.

With this background, the general aim of this project is to increase the knowledge on the influence of nutritional/lifestyle interventions in obese patients with NAFLD, as well as contribute to identify non-invasive biomarkers/scores to early diagnosis of this pathology in future obese people.

DETAILED DESCRIPTION:
This project is framed within the promotion of health and lifestyles and, specifically, in liver disorder linked to obesity (FLiO: Fatty Liver in Obesity).

The investigation addresses a randomized, parallel, long-term personalized nutritional intervention with two strategies: 1) Control diet based on American Heart Association (AHA); 2) Fatty Liver in Obesity (FLiO) diet based on previous results (RESMENA project).The diet is based on macronutrient distribution, quality and quantity, and is characterized by a low glycemic load, high adherence to the Mediterranean diet and a high antioxidant capacity, with the inclusion of anti-inflammatory foods. It also takes into account the distribution of food throughout the day, number of meals, portion sizes, timing of meal, individual needs, dietary behavior (behavioral therapy: eat slowly, teach what to buy, what to eat, when to eat). The participants are instructed to follow this strategy. This strategy (RESMENA) was even more effective than AHA after 6 months follow-up, in terms of significant reduction of abdominal fat and blood glucose level. In addition, this diet had beneficial effects for participants who were obese and had values of altered glucose, reducing significantly in RESMENA participants LDL-oxidized marker. These results are very important to apply in the present investigation since that patients with NAFLD are commonly insulin resistant.

Both strategies were designed within a hypocaloric dietary pattern (-30%) in order to achieve the American Association for the Study of Liver Diseases (AASLD) recommendations for the management of non-alcoholic liver disease (loss of at least 3-5% of body weight appears necessary to improve steatosis, but a greater weight loss, up to 10%, may be needed to improve necroinflammation). At this time the participants are individually supervised and encouraged to follow with the dietary planning instructions assigned. Furthermore, at baseline, 6, 12 and 24 months anticipated variables are obtained. Both dietary groups receive routine control (weight, body composition, strategy adherence) and dietary advice daily by phone (if they need help) and face to face at the time of routine control.

In order to get a integral lifestyle intervention, all participants will be encouraged to follow a healthy lifestyle. Thus, physical activity will be recorded in each dietary group.

The specific tasks:

1. To recruit and select patients with the adequate characteristics to validate the conclusions reached.
2. To develop and adequately transmit to each patient a personalized strategy according to the group randomly assigned ( AASLD vs FLiO strategy).
3. To check the degree of adherence to the strategy set by regular monitoring: semiquantitative questionnaires of food consumption frequency, pedometers, accelerometers, weight control, satiety.
4. To assess the effect of each strategy on body composition (weight, waist circumference, body fat, muscle mass, bone mineral density), physical status, general biochemistry (lipid profile, glycaemic profile, albumin, blood count, transaminases), specific biomarkers/metabolites in blood or urine (inflammation, oxidative stress, liver damage, appetite, psychological status), quality of life and related factors (anxiety, depression and sleep).
5. To check the evolution of the liver damage, using non-invasive techniques (ultrasound, elastography and magnetic resonance imaging (MRI), metabolomics analysis) and calculating different validated liver scores from the data obtained with each strategy.
6. To compare the effectiveness of strategies, considering not only the ability to decrease body fat, but also other risk factors present in the NAFLD patient such as insulin resistance and cardiovascular risk, which will result in improvement of liver damage.
7. To analyze SNPs (DNA from oral epithelial cells) and the association with NAFLD (diagnosis and response to the strategies).
8. To study gene expression (mRNAs) and microRNAs in white blood cells for identifying biomarkers of diagnosis and response to dietary strategy.
9. To analyze gene DNA methylation patterns in white blood cells for identifying biomarkers of diagnosis and response to dietary strategy.
10. To describe the intestinal microbiota composition by 16s sequencing at baseline and after nutritional intervention for diagnosis and response.

ELIGIBILITY:
Inclusion Criteria:

* Overweight or obese
* Diagnosis of NAFLD
* Age: 30-80 years
* Female / Male

Exclusion Criteria:

* Known liver disease (other than NAFLD)
* Abuse of alcohol (>21 and >14 units of alcohol a week for men and women, respectively, eg 1 unit = 125 mL of wine);
* Drug treatments: immunosuppressants, cytotoxic agents, systemic corticosteroids, agents potentially causing fatty liver disease or abnormal liver tests or weight modifiers
* Active cancer or a history of malignancy in the last 5 years
* Problems of massive edemas
* Obesity known endocrine origin (except treated hypothyroidism)
* Surgical procedure for weight loss
* ≥ 3kg weight loss in the last 3 months
* Severe psychiatric disorders
* Lack of autonomy or inability to follow the diet (including food allergies or intolerances) or/and lifestyle recommendations as well as to follow scheduled visits.
* Consumption of any type of food supplements (antioxidants, prebiotics, probiotics, etc.)

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-06 (Actual); Primary Completion 2017-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Weight at 6 months | Baseline and 6 months
  Weight will be measured by a digital scale
Change from 6 month Weight at 12 months | 6 months and 12 months
  Weight will be measured by a digital scale
Change from Baseline Weight at 12 months | Baseline and 12 months
  Weight will be measured by a digital scale

SECONDARY OUTCOMES:
Change from Baseline Body fat at 6 months | Baseline and 6 months
  Fat mass will be measured by Dual X-ray absorptiometry
Change from 6 month Body fat at 12 months | 6 months and 12 months
  Fat mass will be measured by Dual X-ray absorptiometry
Change from Baseline Body fat at 12 months | Baseline and 12 months
  Fat mass will be measured by Dual X-ray absorptiometry
Change from Baseline Waist circumference at 6 months | Baseline and 6 months
  Waist circumference will be measured with a tape measure
Change from 6 month Waist circumference at 12 months | 6 months and 12 months
  Waist circumference will be measured with a tape measure
Change from Baseline Waist circumference at 12 months | Baseline and 12 months
  Waist circumference will be measured with a tape measure
Change from Baseline handgrip strength at 6 months | Baseline and 6 months
  Handgrip strength will be measured with a dynamometer
Change from 6 month handgrip strength at 12 months | 6 months and 12 months
  Handgrip strength will be measured with a dynamometer
Change from Baseline handgrip strength at 12 months | Baseline and 12 months
  Handgrip strength will be measured with a dynamometer
Change from Baseline Systolic blood pressure at 6 months | Baseline and 6 months
  Systolic blood pressure will be measured with a sphygmomanometer
Change from 6 month Systolic blood pressure at 12 months | 6 months and 12 months
  Systolic blood pressure will be measured with a sphygmomanometer
Change from Baseline Systolic blood pressure at 12 months | Baseline and 12 months
  Systolic blood pressure will be measured with a sphygmomanometer
Change from Baseline Diastolic blood pressure at 6 months | Baseline and 6 months
  Diastolic blood pressure will be measured with a sphygmomanometer
Change from 6 month Diastolic blood pressure at 12 months | 6 months and 12 months
  Diastolic blood pressure will be measured with a sphygmomanometer
Change from Baseline Diastolic blood pressure at 12 months | Baseline and 12 months
  Diastolic blood pressure will be measured with a sphygmomanometer
Change from Baseline lipid metabolism at 6 months | Baseline and 6 months
  Serum free fatty acids, triglycerides, total cholesterol, LDL cholesterol and HDL cholesterol concentrations will be measured in a fasting state
Change from 6 month lipid metabolism at 12 months | 6 months and 12 months
  Serum free fatty acids, triglycerides, total cholesterol, LDL cholesterol and HDL cholesterol concentrations will be measured in a fasting state
Change from Baseline lipid metabolism at 12 months | Baseline and 12 months
  Serum free fatty acids, triglycerides, total cholesterol, LDL cholesterol and HDL cholesterol concentrations will be measured in a fasting state
Change from Baseline uric acid concentration at 6 months | Baseline and 6 months
  Serum uric acid will be measured in a fasting state
Change from 6 month uric acid concentration at 12 months | 6 months and 12 months
  Serum uric acid will be measured in a fasting state
Change from Baseline uric acid concentration at 12 months | Baseline and 12 months
  Serum uric acid will be measured in a fasting state
Change from Baseline homocysteine concentration at 6 months | Baseline and 6 months
  Serum homocysteine will be measured in a fasting state
Change from 6 month homocysteine concentration at 12 months | 6 months and 12 months
  Serum homocysteine will be measured in a fasting state
Change from Baseline homocysteine concentration at 12 months | Baseline and 12 months
  Serum homocysteine will be measured in a fasting state
Change from Baseline glucose metabolism at 6 months | Baseline and 6 months
  Serum glucose levels will be measured in a fasting state
Change from 6 month glucose metabolism at 12 months | 6 months and 12 months
  Serum glucose levels will be measured in a fasting state
Change from Baseline glucose metabolism at 12 months | Baseline and 12 months
  Serum glucose levels will be measured in a fasting state
Change from Baseline insulin concentration at 6 months | Baseline and 6 months
  Serum insulin levels will be measured in a fasting state
Change from 6 month insulin concentration at 12 months | 6 months and 12 months
  Serum insulin levels will be measured in a fasting state
Change from Baseline insulin concentration at 12 months | Baseline and 12 months
  Serum insulin levels will be measured in a fasting state
Change from Baseline Hemoglobin A1c concentration at 6 months | Baseline and 6 months
  Serum Hemoglobin A1c will be measured in a fasting state
Change from 6 month Hemoglobin A1c concentration at 12 months | 6 months and 12 months
  Serum Hemoglobin A1c will be measured in a fasting state
Change from Baseline Hemoglobin A1c concentration at 12 months | Baseline and 12 months
  Serum Hemoglobin A1c will be measured in a fasting state
Change from Baseline liver function at 6 months | Baseline and 12 months
  Serum aspartate aminotransferase, alanine aminotransferase, gamma-glutamyltransferase, total bilirubin, direct bilirubin, alkaline phosphatase, creatinine, total protein, albumin, prothrombin will be measured in a fasting state
Change from 6 month liver function at 12 months | 6 months and 12 months
  Serum aspartate aminotransferase, alanine aminotransferase, gamma-glutamyltransferase, total bilirubin, direct bilirubin, alkaline phosphatase, creatinine, total protein, albumin, prothrombin will be measured in a fasting state
Change from Baseline liver function at 12 months | Baseline and 12 months
  Serum aspartate aminotransferase, alanine aminotransferase, gamma-glutamyltransferase, total bilirubin, direct bilirubin, alkaline phosphatase, creatinine, total protein, albumin, prothrombin will be measured in a fasting state
Change from Baseline fibroblast growth factor 21 (FGF21) concentration at 6 months | Baseline and 6 months
  Plasma FGF21 is a specific biomarker of NAFLD and will be measured in a fasting state
Change from 6 month fibroblast growth factor 21 (FGF21) concentration at 12 months | 6 months and 12 months
  Plasma FGF21 is a specific biomarker of NAFLD and will be measured in a fasting state
Change from Baseline fibroblast growth factor 21 (FGF21) concentration at 12 months | Baseline and 12 months
  Plasma FGF21 is a specific biomarker of NAFLD and will be measured in a fasting state
Change from Baseline cytokeratin-18 (CK18) concentration at 6 months | Baseline and 6 months
  Plasma CK18 is a specific biomarker of NAFLD and will be measured in a fasting state
Change from 6 month cytokeratin-18 (CK18) concentration at 12 months | 6 months and 12 months
  Plasma CK18 is a specific biomarker of NAFLD and will be measured in a fasting state
Change from Baseline cytokeratin-18 (CK18) concentration at 12 months | Baseline and 12 months
  Plasma CK18 is a specific biomarker of NAFLD and will be measured in a fasting state
Change from Baseline C-reactive protein (CRP) concentration at 6 months | Baseline and 6 months
  Plasma CRP will be assessed to determine inflammatory status
Change from 6 month C-reactive protein (CRP) concentration at 12 months | 6 months and 12 months
  Plasma CRP will be assessed to determine inflammatory status
Change from Baseline C-reactive protein (CRP) concentration at 12 months | Baseline and 12 months
  Plasma CRP will be assessed to determine inflammatory status
Change from Baseline interleukin 6 (IL-6) concentration at 6 months | Baseline and 6 months
  Plasma IL-6 will be assessed to determine inflammatory status
Change from 6 month interleukin 6 (IL-6) concentration at 12 months | 6 months and 12 months
  Plasma IL-6 will be assessed to determine inflammatory status
Change from Baseline interleukin 6 (IL-6) concentration at 12 months | Baseline and 12 months
  Plasma IL-6 will be assessed to determine inflammatory status
Change from Baseline tumor necrosis factor-α (TNFα) concentration at 6 months | Baseline and 6 months
  Plasma TNF-alpha will be assessed to determine inflammatory status
Change from 6 month tumor necrosis factor-α (TNFα) concentration at 12 months | 6 months and 12 months
  Plasma TNF-alpha will be assessed to determine inflammatory status
Change from Baseline tumor necrosis factor-α (TNFα) concentration at 12 months | Baseline and 12 months
  Plasma TNF-alpha will be assessed to determine inflammatory status
Change from Baseline leptin concentration at 6 months | Baseline and 6 months
  Plasma leptin will be assessed to determine inflammatory status
Change from 6 month leptin concentration at 12 months | 6 months and 12 months
  Plasma leptin will be assessed to determine inflammatory status
Change from Baseline leptin concentration at 12 months | Baseline and 12 months
  Plasma leptin will be assessed to determine inflammatory status
Change from Baseline adiponectin concentration at 6 months | Baseline and 6 months
  Plasma leptin will be assessed to determine inflammatory status
Change from 6 month adiponectin concentration at 12 months | Baseline and 12 months
  Plasma adiponectin will be assessed to determine inflammatory status
Change from Baseline adiponectin concentration at 12 months | Baseline and 12 months
  Plasma adiponectin will be assessed to determine inflammatory status
Change from Baseline LDL-oxidized concentration at 6 months | Baseline and 6 months
  LDL-ox will be assessed to determine oxidative status
Change from 6 month LDL-oxidized concentration at 12 months | 6 months and 12 months
  LDL-ox will be assessed to determine oxidative status
Change from Baseline LDL-oxidized concentration at 12 months | Baseline and 12 months
  LDL-ox will be assessed to determine oxidative status
Change from Baseline Malondialdehyde concentration at 6 months | Baseline and 6 months
  Plasma malondialdehyde will be assessed to determine oxidative status
Change from 6 month Malondialdehyde concentration at 12 months | 6 months and 12 months
  Plasma malondialdehyde will be assessed to determine oxidative status
Change from Baseline Malondialdehyde concentration at 12 months | Baseline and 12 months
  Plasma malondialdehyde will be assessed to determine oxidative status
Change from Baseline plasma antioxidant capacity at 6 months | Baseline and 6 months
  Plasma antioxidant capacity will be assessed by measuring the ferric reducing ability of plasma (FRAP)
Change from 6 month plasma antioxidant capacity at 12 months | 6 months and 12 months
  Plasma antioxidant capacity will be assessed by measuring the ferric reducing ability of plasma (FRAP)
Change from Baseline plasma antioxidant capacity at 12 months | Baseline and 12 months
  Plasma antioxidant capacity will be assessed by measuring the ferric reducing ability of plasma (FRAP)
Change from Baseline Hepatic echography at 6 months | Baseline and 6 months
  Echography will be carried out to analyze liver steatosis
Change from 6 month Hepatic echography at 12 months | 6 months and 12 months
  Echography will be carried out to analyze liver steatosis
Change from Baseline Hepatic echography at 12 months | Baseline and 12 months
  Echography will be carried out to analyze liver steatosis
Change from Baseline Hepatic elastography at 6 months | Baseline and 6 months
  Elastography will be carried out to analyze liver fibrosis
Change from 6 month Hepatic elastography at 12 months | 6 months and 12 months
  Elastography will be carried out to analyze liver fibrosis
Change from Baseline Hepatic elastography at 12 months | Baseline and 12 months
  Elastography will be carried out to analyze liver fibrosis
Change from Baseline Hepatic Magnetic Resonance Imaging at 6 months | Baseline and 6 months
  Magnetic Resonance Imaging will be carried out to analyze liver status
Change from 6 month Hepatic Magnetic Resonance Imaging at 12 months | 6 months and 12 months
  Magnetic Resonance Imaging will be carried out to analyze liver status
Change from Baseline Hepatic Magnetic Resonance Imaging at 12 months | Baseline and 12 months
  Magnetic Resonance Imaging will be carried out to analyze liver status
Change from Baseline White blood cell count at 6 months | Baseline and 6 months
  White blood cell count includes: Leucocytes, Neutrophils, Lymphocytes, Monocytes, Eosinophil, Basophils.
Change from 6 month White blood cell count at 12 months | 6 months and 12 months
  White blood cell count includes: Leucocytes, Neutrophils, Lymphocytes, Monocytes, Eosinophil, Basophils.
Change from Baseline White blood cell count at 12 months | Baseline and 12 months
  White blood cell count includes: Leucocytes, Neutrophils, Lymphocytes, Monocytes, Eosinophil, Basophils.
Change from Baseline blood rheological properties at 6 months | Baseline and 6 months
  Red blood cell count, hematocrit, mean corpuscular volume, mean corpuscular hemoglobin, mean corpuscular hemoglobin concentration, red cell distribution width, platelet count, platelet distribution width, mean platelet volume, plateletcrit
Change from 6 month blood rheological properties at 12 months | 6 months and 12 months
  Red blood cell count, hematocrit, mean corpuscular volume, mean corpuscular hemoglobin, mean corpuscular hemoglobin concentration, red cell distribution width, platelet count, platelet distribution width, mean platelet volume, plateletcrit
Change from Baseline blood rheological properties at 12 months | Baseline and 12 months
  Red blood cell count, hematocrit, mean corpuscular volume, mean corpuscular hemoglobin, mean corpuscular hemoglobin concentration, red cell distribution width, platelet count, platelet distribution width, mean platelet volume, plateletcrit
Change from Baseline Physical activity level at 6 months | Baseline and 6 months
  Physical activity will be assessed by accelerometers
Change from 6 months Physical activity level at 12 months | 6 months and 12 months
  Physical activity will be assessed accelerometers
Change from Baseline Physical activity level at 12 months | Baseline and 12 months
  Physical activity will be assessed by accelerometers
Change from Baseline Minnesota Physical Activity test at 6 months | Baseline and 6 months
  Physical activity assessed by Minnesota Physical Activity test
Change from 6 month Minnesota Physical Activity test at 12 months | 6 months and 12 months
  Physical activity assessed by Minnesota Physical Activity test
Change from Baseline Minnesota Physical Activity test at 12 months | Baseline and 12 months
  Physical activity assessed by Minnesota Physical Activity test
Change from Baseline number of steps at 6 months | Baseline and 6 months
  Physical activity assessed by Pedometers
Change from 6 month number of steps at 12 months | 6 months and 12 months
  Physical activity assessed by Pedometers
Change from Baseline number of steps at 12 months | Baseline and 12 months
  Physical activity assessed by Pedometers
Change from Baseline chair test at 6 months | Baseline and 6 months
  Physical activity assessed by the chair test
Change from 6 month chair test at 12 months | 6 months and 12 months
  Physical activity assessed by the chair test
Change from Baseline chair test at 12 months | Baseline and 12 months
  Physical activity assessed by the chair test
Change from Baseline sleep quality at 6 months | Baseline and 12 months
  Sleep information will be assessed by the Pittsburgh Sleep Quality Index
Change from 6 month sleep quality at 12 months | 6 months and 12 months
  Sleep information will be assessed by the Pittsburgh Sleep Quality Index
Change from Baseline sleep quality at 12 months | Baseline and 12 months
  Sleep information will be assessed by the Pittsburgh Sleep Quality Index
Change from Baseline Depressive symptoms at 6 months | Baseline and 6 months
  Depressive symptoms will be assessed by the Beck Depression Inventory (BDI)
Change from 6 month Depressive symptoms at 12 months | 6 months and 12 months
  Depressive symptoms will be assessed by the Beck Depression Inventory (BDI)
Change from Baseline Depressive symptoms at 12 months | Baseline and 12 months
  Depressive symptoms will be assessed by the Beck Depression Inventory (BDI)
Change from Baseline Anxiety symptoms at 6 months | Baseline and 6 months
  Anxiety symptoms will be assessed by State Anxiety test (STAI)
Change from 6 month Anxiety symptoms at 12 months | 6 months and 12 months
  Anxiety symptoms will be assessed by State Anxiety test (STAI)
Change from Baseline Anxiety symptoms at 12 months | Baseline and 12 months
  Anxiety symptoms will be assessed by State Anxiety test (STAI)
Single Nucleotide polymorphisms (SNPs) | Baseline
  Single nucleotide polymorphisms will be determined by Genomic DNA from oral epithelial cells
Change from Baseline DNA methylation at 6 months | Baseline and 6 months
  Epigenetics will be assessed by changes in DNA methylation of genes related with NAFLD development
Change from 6 month DNA methylation at 12 months | 6 months and 12 months
  Epigenetics will be assessed by changes in DNA methylation of genes related with NAFLD development
Change from Baseline DNA methylation at 12 months | Baseline and 12 months
  Epigenetics will be assessed by changes in DNA methylation of genes related with NAFLD development
Change from Baseline microRNAs at 6 months | Baseline and 6 months
  Transcriptomic will be assessed by changes in miRNAs
Change from 6 month microRNAs at 12 months | 6 months and 12 months
  Transcriptomic will be assessed by changes in miRNAs
Change from Baseline microRNAs at 12 months | Baseline and 12 months
  Transcriptomic will be assessed by changes in miRNAs
Change from Baseline Gut microbiota composition at 6 months | Baseline and 6 months
  Gut microbiota composition will be analyzed
Change from 6 month Gut microbiota composition at 12 month | 6 months and 12 months
  Gut microbiota composition will be analyzed
Change from Baseline Gut microbiota composition at 12 month | Baseline and 12 months
  Gut microbiota composition will be analyzed
Change from Baseline metabolites composition of urine at 6 months | Baseline and 6 months
  Metabolites composition of urine will be analyzed
Change from 6 month metabolites composition of urine at 12 months | 6 months and 12 months
  Metabolites composition of urine will be analyzed
Change from Baseline metabolites composition of urine at 12 months | Baseline and 12 months
  Metabolites composition of urine will be analyzed
Change from Baseline metabolites composition of serum at 6 months | Baseline and 6 months
  Metabolites composition of serum will be analyzed
Change from 6 month metabolites composition of serum at 12 months | 6 months and 12 months
  Metabolites composition of serum will be analyzed
Change from Baseline metabolites composition of serum at 12 months | Baseline and 12 months
  Metabolites composition of serum will be analyzed
Change from Baseline dietary intake at 6 months | Baseline and 6 months
  Dietary intake will be assessed by means of food frequency questionnaire
Change from 6 month dietary intake at 12 months | 6 months and 12 months
  Dietary intake will be assessed by means of food frequency questionnaire
Change from Baseline dietary intake at 12 months | Baseline and 12 months
  Dietary intake will be assessed by means of food frequency questionnaire
Assessment of dietary adherence at Baseline | Baseline
  Dietary adherence will be assessed by means of 3 day weighed food records
Assessment of dietary adherence at 6 months | 6 months
  Dietary adherence will be assessed by means of 3 day weighed food records
Assessment of dietary adherence at 12 months | 12 months
  Dietary adherence will be assessed by means of 3 day weighed food records
Change from Baseline satiety index at 6 months | Baseline and 6 months
  Satiety index/appetite will be assessed by using the 100 mm Visual Analogue Scale
Change from 6 month satiety index at 12 months | 6 months and 12 months
  Satiety index/appetite will be assessed by using the 100 mm Visual Analogue Scale
Change from Baseline satiety index at 12 months | Baseline and 12 months
  Satiety index/appetite will be assessed by using the 100 mm Visual Analogue Scale
Change from Baseline life quality index at 6 months | Baseline and 6 months
  Life quality index will be assessed by means of the Short Form 36 (SF-36) questionnaire
Change from 6 month life quality index at 12 months | 6 months and 12 months
  Life quality index will be assessed by means of the Short Form 36 (SF-36) questionnaire
Change from Baseline life quality index at 12 months | Baseline and 12 months
  Life quality index will be assessed by means of the Short Form 36 (SF-36) questionnaire
Change from Baseline Ghrelin concentration at 6 months | Baseline and 6 months
  Serum Active Ghrelin will be determined to assess satiety
Change from 6 month Ghrelin concentration at 12 months | 6 months and 12 months
  Serum Active Ghrelin will be determined to assess satiety
Change from Baseline Ghrelin concentration at 12 months | Baseline and 12 months
  Serum Active Ghrelin will be determined to assess satiety
Change from Baseline glucagon-like peptide-1 (GLP-1) concentration at 6 months | Baseline and 6 months
  Serum active glucagon-like peptide-1 will be determined to assess satiety
Change from 6 month glucagon-like peptide-1 (GLP-1) concentration at 12 months | 6 months and 12 months
  Serum active glucagon-like peptide-1 will be determined to assess satiety
Change from Baseline glucagon-like peptide-1 (GLP-1) concentration at 12 months | Baseline and 12 months
  Serum active glucagon-like peptide-1 will be determined to assess satiety
Change from Baseline Dopamine concentration at 6 months | Baseline and 6 months
  Peripheral Dopamine concentration will be analysed using high-performance liquid chromatography (HPLC)
Change from 6 month Dopamine concentration at 12 months | 6 months and 12 months
  Peripheral Dopamine concentration will be analysed using high-performance liquid chromatography (HPLC)
Change from Baseline Dopamine concentration at 12 months | Baseline and 12 months
  Peripheral Dopamine concentration will be analysed using high-performance liquid chromatography (HPLC)
Change from Baseline Dopac concentration at 6 months | Baseline and 6 months
  Peripheral Dopac concentration will be analysed using high-performance liquid chromatography (HPLC)
Change from 6 month Dopac concentration at 12 months | 6 months and 12 months
  Peripheral Dopac concentration will be analysed using high-performance liquid chromatography (HPLC)
Change from Baseline Dopac concentration at 12 months | Baseline and 12 months
  Peripheral Dopac concentration will be analysed using high-performance liquid chromatography (HPLC)
Change from Baseline Serotonin (5-HT) concentration at 6 months | Baseline and 6 months
  Peripheral Serotonin concentration will be analysed using high-performance liquid chromatography (HPLC)
Change from 6 month Serotonin (5-HT) concentration at 12 months | 6 months and 12 months
  Peripheral Serotonin concentration will be analysed using high-performance liquid chromatography (HPLC)
Change from Baseline Serotonin (5-HT) concentration at 12 months | Baseline and 12 months
  Peripheral Serotonin concentration will be analysed using high-performance liquid chromatography (HPLC)
Change from Baseline Noradrenaline concentration at 6 months | Baseline and 6 months
  Peripheral Noradrenaline concentration will be analysed using high-performance liquid chromatography (HPLC)
Change from 6 month Noradrenaline concentration at 12 months | 6 months and 12 months
  Peripheral Noradrenaline concentration will be analysed using high-performance liquid chromatography (HPLC)
Change from Baseline Noradrenaline concentration at 12 months | Baseline and 12 months
  Peripheral Noradrenaline concentration will be analysed using high-performance liquid chromatography (HPLC)
Change from Baseline 5-hydroxyindoleacetic acetic (5-HIAAC) concentration at 6 months | Baseline and 6 months
  Peripheral 5-hydroxyindoleacetic acetic concentration will be analysed using high-performance liquid chromatography (HPLC)
Change from 6 month 5-hydroxyindoleacetic acetic (5-HIAAC) concentration at 12 months | 6 months and 12 months
  Peripheral 5-hydroxyindoleacetic acetic concentration will be analysed using high-performance liquid chromatography (HPLC)
Change from Baseline 5-hydroxyindoleacetic acetic (5-HIAAC) concentration at 12 months | Baseline and 12 months
  Peripheral 5-hydroxyindoleacetic acetic concentration will be analysed using high-performance liquid chromatography (HPLC)

CONTACTS AND LOCATIONS:
Overall Officials: M. Angeles Zulet, PhD, Principal Investigator — Centre for Nutrition Research, University of Navarra. CIBER Obesity and Physiopathology of Nutrition (CIBERobn), Institute of Health Carlos III, Madrid, Spain; J. Alfredo Martínez, MD, PhD, Study Director — Centre for Nutrition Research, University of Navarra. CIBER Obesity and Physiopathology of Nutrition (CIBERobn), Institute of Health Carlos III, Madrid, Spain; Itziar Abete, PhD, Study Director — Centre for Nutrition Research, University of Navarra. CIBER Obesity and Physiopathology of Nutrition (CIBERobn), Institute of Health Carlos III, Madrid, Spain; Fermín I Milagro, PhD, Study Chair — Centre for Nutrition Research, University of Navarra. CIBER Obesity and Physiopathology of Nutrition (CIBERobn), Institute of Health Carlos III, Madrid, Spain; J. Ignacio Riezu, PhD, Study Chair — Centre for Nutrition Research, University of Navarra.; Mariana Elorz, MD, Study Chair — Clínica Universidad de Navarra; J. Ignacio Herrero, PhD, Study Chair — Clinica Universidad de Navarra; Jorge Quiroga, PhD, Study Chair — Clinica Universidad de Navarra; Alberto Benito, PhD, Study Chair — Clinica Universidad de Navarra; Carmen Fuertes, Study Chair — Clinica Universidad de Navarra; Santiago Navas, PhD, Study Chair — Centre for Nutrition Research, University of Navarra. CIBER Obesity and Physiopathology of Nutrition (CIBERobn), Institute of Health Carlos III, Madrid, Spain; Eva Almirón, PhD, Study Chair — Centre for Nutrition Research, University of Navarra.; Berta Araceli Marín, Study Chair — University of Navarra; Irene Cantero, Study Chair — University of Navarra; Maria Vanessa Bullon, Study Chair — University of Navarra; Blanca Martínez de Morentín, MD, Study Chair — University of Navarra; Salomé Pérez, Study Chair — University of Navarra; Veronica Ciaurriz, Study Chair — University of Navarra; Ana Martínez, MD, Study Chair — Complejo Hospitalario de Navarra; Juan Uriz, PhD, Study Chair — Complejo Hospitalario de Navarra; María Pilar Huarte, PhD, Study Chair — Complejo Hospitalario de Navarra; J. Ignacio Monreal, MD, PhD, Study Chair — Clinica Universidad de Navarra
Locations (1):
- Centre for Nutrition Research, University of Navarra, Pamplona, Navarre, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Abd El-Kader SM, El-Den Ashmawy EM. Non-alcoholic fatty liver disease: The diagnosis and management. World J Hepatol. 2015 Apr 28;7(6):846-58. doi: 10.4254/wjh.v7.i6.846. PMID 25937862
- [Background] de la Iglesia R, Lopez-Legarrea P, Abete I, Bondia-Pons I, Navas-Carretero S, Forga L, Martinez JA, Zulet MA. A new dietary strategy for long-term treatment of the metabolic syndrome is compared with the American Heart Association (AHA) guidelines: the MEtabolic Syndrome REduction in NAvarra (RESMENA) project. Br J Nutr. 2014 Feb;111(4):643-52. doi: 10.1017/S0007114513002778. Epub 2013 Aug 23. PMID 23968597
- [Background] de la Iglesia R, Lopez-Legarrea P, Celada P, Sanchez-Muniz FJ, Martinez JA, Zulet MA. Beneficial effects of the RESMENA dietary pattern on oxidative stress in patients suffering from metabolic syndrome with hyperglycemia are associated to dietary TAC and fruit consumption. Int J Mol Sci. 2013 Mar 27;14(4):6903-19. doi: 10.3390/ijms14046903. PMID 23535332
- [Background] Lopez-Legarrea P, de la Iglesia R, Abete I, Bondia-Pons I, Navas-Carretero S, Forga L, Martinez JA, Zulet MA. Short-term role of the dietary total antioxidant capacity in two hypocaloric regimes on obese with metabolic syndrome symptoms: the RESMENA randomized controlled trial. Nutr Metab (Lond). 2013 Feb 13;10(1):22. doi: 10.1186/1743-7075-10-22. PMID 23406163
- [Background] Yasutake K, Kohjima M, Kotoh K, Nakashima M, Nakamuta M, Enjoji M. Dietary habits and behaviors associated with nonalcoholic fatty liver disease. World J Gastroenterol. 2014 Feb 21;20(7):1756-67. doi: 10.3748/wjg.v20.i7.1756. PMID 24587653
- [Result] Chalasani N, Younossi Z, Lavine JE, Diehl AM, Brunt EM, Cusi K, Charlton M, Sanyal AJ; American Gastroenterological Association; American Association for the Study of Liver Diseases; American College of Gastroenterologyh. The diagnosis and management of non-alcoholic fatty liver disease: practice guideline by the American Gastroenterological Association, American Association for the Study of Liver Diseases, and American College of Gastroenterology. Gastroenterology. 2012 Jun;142(7):1592-609. doi: 10.1053/j.gastro.2012.04.001. Epub 2012 May 15. No abstract available. PMID 22656328
- [Derived] Tobaruela-Resola AL, Riezu-Boj JI, Milagro FI, Mogna-Pelaez P, Herrero JI, Elorz M, Benito-Boillos A, Tur JA, Martinez JA, Abete I, Zulet MA. Circulating microRNA panels in subjects with metabolic dysfunction-associated steatotic liver disease after following a 2-year dietary intervention. J Endocrinol Invest. 2025 Apr;48(4):987-1003. doi: 10.1007/s40618-024-02499-9. Epub 2024 Nov 16. PMID 39549213
- [Derived] Mogna-Pelaez P, Riezu-Boj JI, Milagro FI, Herrero JI, Elorz M, Benito-Boillos A, Tobaruela-Resola AL, Tur JA, Martinez JA, Abete I, Zulet MA. Inflammatory markers as diagnostic and precision nutrition tools for metabolic dysfunction-associated steatotic liver disease: Results from the Fatty Liver in Obesity trial. Clin Nutr. 2024 Jul;43(7):1770-1781. doi: 10.1016/j.clnu.2024.05.042. Epub 2024 May 31. PMID 38861890
- [Derived] Marin-Alejandre BA, Cantero I, Perez-Diaz-Del-Campo N, Monreal JI, Elorz M, Herrero JI, Benito-Boillos A, Quiroga J, Martinez-Echeverria A, Uriz-Otano JI, Huarte-Muniesa MP, Tur JA, Martinez JA, Abete I, Zulet MA. Effects of two personalized dietary strategies during a 2-year intervention in subjects with nonalcoholic fatty liver disease: A randomized trial. Liver Int. 2021 Jul;41(7):1532-1544. doi: 10.1111/liv.14818. Epub 2021 Mar 1. PMID 33550706
- [Derived] Perez-Diaz-Del-Campo N, Marin-Alejandre BA, Cantero I, Monreal JI, Elorz M, Herrero JI, Benito-Boillos A, Riezu-Boj JI, Milagro FI, Tur JA, Martinez JA, Abete I, Zulet MA. Differential response to a 6-month energy-restricted treatment depending on SH2B1 rs7359397 variant in NAFLD subjects: Fatty Liver in Obesity (FLiO) Study. Eur J Nutr. 2021 Sep;60(6):3043-3057. doi: 10.1007/s00394-020-02476-x. Epub 2021 Jan 20. PMID 33474638
- [Derived] Galarregui C, Cantero I, Marin-Alejandre BA, Monreal JI, Elorz M, Benito-Boillos A, Herrero JI, de la O V, Ruiz-Canela M, Hermsdorff HHM, Bressan J, Tur JA, Martinez JA, Zulet MA, Abete I. Dietary intake of specific amino acids and liver status in subjects with nonalcoholic fatty liver disease: fatty liver in obesity (FLiO) study. Eur J Nutr. 2021 Jun;60(4):1769-1780. doi: 10.1007/s00394-020-02370-6. Epub 2020 Aug 28. PMID 32857176
- [Derived] Cantero I, Elorz M, Abete I, Marin BA, Herrero JI, Monreal JI, Benito A, Quiroga J, Martinez A, Huarte MP, Uriz-Otano JI, Tur JA, Kearney J, Martinez JA, Zulet MA. Ultrasound/Elastography techniques, lipidomic and blood markers compared to Magnetic Resonance Imaging in non-alcoholic fatty liver disease adults. Int J Med Sci. 2019 Jan 1;16(1):75-83. doi: 10.7150/ijms.28044. eCollection 2019. PMID 30662331